CLINICAL TRIAL: NCT06594549
Title: Sleep Health, Workplace Stress and Wellbeing in NUS Staff: the NUS1000 Staff Edition Study
Acronym: NUS1000SE
Status: Not yet recruiting | Type: Observational
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Michael W.L. Chee, Professor, National University of Singapore
Other Study IDs: NUS1000 staff edition
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Life Experiences
Keywords: Employee; Sleep; Wellbeing; Stress; Cardiovascular; Workplace

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Staff: NUS Staff

SUMMARY:
Workplace stress can significantly affect workers sleep, physical health and mental wellbeing. Recognizing and characterizing obstacles to healthy sleep patterns in office workers can help identify targets for corporate interventions that improve productivity and workplace wellbeing. Following the investigator's experience with the NUS1000 study in 1st year students conducted in Aug-Dec 2023, the investigators will now track daily sleep, wellbeing and time-use in NUS staff for 1 year in the present study. These data will reveal work-related stressors that impact daily sleep and mood. In addition, the investigators will investigate whether daily sleep and stress are associated with cardiovascular health in this middle-age cohort.

DETAILED DESCRIPTION:
The investigators aim to answer the following questions using a combination of objective sleep tracking (Oura ring), smartphone-based questionnaires (EMA), passive tracking of interactions on smartphones (Quantactions) and one-time arterial stiffness measures (SphygmoCor).

1. Identify obstacles to healthy sleep patterns in NUS staff 1.1) How do staff sleep, in terms of duration, timing, regularity and napping behaviour? 1.2) What is the gulf between sleep aspiration and attained sleep? 1.3) What are self-perceived obstacles to achieving better sleep? 1.4) What activities potentially displace time for sleep?
2. Understand inter-relationships between sleep, workplace stressors and wellbeing outcomes 2.1) How is sleep is modulated over the year? 2.2) How do work patterns (e.g., after-hours/vacation emails) correlate with sleep, physical activity, subjective wellbeing, physiological markers of stress? 2.3) How do work, social, status stress and other life events contribute to sleep, wellbeing and subjective perceptions of work productivity?
3. Examine the association between sleep, workplace stress, mental health, cardiovascular risks in middle-aged cohort 3.1) How do daily sleep, work place events and acute/chronic stress contribute to cardiovascular health atmiddle age? 3.2) How is subjective wellbeing associated with objective cardiovascular wellbeing?
4. Examine the effects of any structural organizational efforts to promote wellbeing on staff sleep and stress

The investigators hypothesize that acute stressors, such as receiving emails after office hours and during vacation periods, will negatively impact sleep duration and regularity, as well as subjective stress rating over a short period. Chronic stressors, such as family care burden and pressure from supervisor, will be associated with longer-term insufficient and irregular sleep. Staff members reporting high chronic stress and frequent acute stress may be more likely to have high cardiovascular and cerebrovascular risks. In general, irregular/short sleep, constant high subjective stress, and frequent routine disruption (i.e., after hours work) will be associated with high cardiovascular risk in middle-aged participants.

ELIGIBILITY:
Inclusion Criteria:

* NUS staff between the age of 35-70 with smartphones operating on Android 8.0 and up, or iOS 14.0 or later

Exclusion Criteria:

Participants will be required to :

1. Have their sleep and physical activity rhythms recorded via wearable sensors, while they continue daily life as usual.
2. Complete periodic questionnaires and short daily surveys on their smartphones.
3. Agree to interactions with their smartphones and NUS e-services (e.g., email) tracked.

Participants who do not agree to have these measures recorded will not be eligible for the study. Shift workers (e.g., security personnel, doctors and nurses), nursing/pregnant woman, and patients with existing sleep/psychological disorders (e.g., insomnia and major depression) will also be excluded.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1000 National University of Singapore staff
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Time-use diary | Across the 1 year study
  Participants will be asked to fill out a time-use diary over 2-week periods every 3 months throughout the follow-up period (Month 1, Month 3, Month 6, Month 9 and Month 12), indicating the activities they engaged in over the past day on the smartphone app.
Blood Pressure | Across the 1 year study
  Blood pressure measures will be taken twice via an Omron blood pressure device.
Arterial Stiffness | Across the 1 year study
  Arterial stiffness will be assessed by SphygmoCor XCEL system (cuff plus tonometer) and pulse wave velocity will be derived.
Height | Across the 1 year study
  Height will be measured by the device linked to the body composition system (cm).
Weight | Across the 1 year study
  Weight will be measured by the device linked to the body composition system (in kg).
Body composition | Across the 1 year study
  Body composition will be assessed by InBody 770 Bioelectrical Impedance Analysis machine.
Smartphone Touchscreen Interactions | Across the 1 year study
  Smartphone taps (number) will be tracked automatically through an EU-GDPR (the European Union's stringent privacy regulation) compliant smartphone app (QuantActions). This application logs human-smartphone screen interactions (e.g., taps, swipes) during regular use by logging a location-specific timestamp for each screen contact, and the name of the active app at that moment. This gives us a readout of phone use, app use, and an implicit measure of alertness (tapping speed). Only timestamps of touchscreen interactions and the associated apps will be recorded. No text, pictures, contacts, or any person identifying information will be collected. Moreover, data will be gathered and stored on the cloud using codes only; names or emails will not be collected.
Sleep time | Across the 1 year study
  The Oura ring is a device worn on the finger which non-invasively records movement, heart rate and temperature to infer sleep and physical activity. Sleep Onset Time, Wake Time, on Workday (weekday) and Free Day (Weekend / vacation) will be recorded for nocturnal sleep and naps.
Sleep duration | Across the 1 year study
  The Oura ring is a device worn on the finger which non-invasively records movement, heart rate and temperature to infer sleep and physical activity. Sleep Duration on Workday (weekday) and Free Day (Weekend / vacation) will be recorded for nocturnal sleep and naps.
Wake after sleep onset | Across the 1 year study
  The Oura ring is a device worn on the finger which non-invasively records movement, heart rate and temperature to infer sleep and physical activity. Wake after Sleep Onset on Workday (weekday) and Free Day (Weekend / vacation) will be recorded.
Sleep regularity | Across the 1 year study
  The Oura ring is a device worn on the finger which non-invasively records movement, heart rate and temperature to infer sleep and physical activity. Sleep Regularity (computed via Std Deviation and Sleep Regularity Index; evaluated over 4 weeks minimally) will be recorded.
Well-being | Across the 1 year study
  Participants input ratings about a rotating set of questions concerning wellbeing daily through a smartphone based app (Z4IP) that has been used in prior studies. This daily assessment can be done anytime between 8pm and 12am each day. Higher scores represent higher levels of well-being.
Self-reported health | Across the 1 year study
  Participants will also be required to complete a subset of health questionnaires every 3 months throughout the follow-up period (Month 1, Month 3,Month 6, Month 9 and Month 12) on the Qualtrics survey platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Yong Loo Lin School of Medicine, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No